## Proprietary of MD Anderson Cancer Center April 24, 2025

NCT05308407

| Date: | |
|-----------------------|-----------|
| Protocol #: _ | 2021-0887 |
| Interviewer Initials: | |

Verbal Script to Obtain Consent for Participation in Protocol 2021-0887, Titled "POWER UP: Participating Online While Exercising to Recover Using Play"

Hello. Is [PATIENT NAME] available?

This is [INTERVIEWER NAME] calling from the Department of Pediatrics Research at The University of Texas MD Anderson Cancer Center. I am calling about a research study that Dr. Keri Schadler is conducting in collaboration with Dr. Michael Roth and Dr. Andy Livingston. The goal of this research study is to get feedback on a new virtual physical activity program.

Would you like to hear more about the study?

- If a participant declines participation, thank them for their time and end the call.
- If the participant agrees to hear more about the study, say:

Do you have any questions before we get started? You can stop me at any time and ask questions.

#### 2. Purpose of the Study

The goal of this research study is to get feedback from adolescents and young adults (or AYAs) on a new virtual physical activity program (called POWER UP) created for AYAs with central nervous system (CNS) tumors.

#### 3. **Study Procedures**

If you agree to take part in this study, you will take part in a focus group interview by video call (using the video conferencing app Zoom) with other AYAs who have CNS tumors. During the focus group, you will be shown the materials that may be used in the POWER UP program. You may also be asked to test some of the active video games that may be used in the program. You will be asked to provide your opinion on the study design and study materials and how to make them more appropriate for AYAs with CNS tumors. Focus groups will be digitally recorded and transcribed (written down). Only audio will be recorded during the focus groups. No videos will be taken of you. After the audio recordings are transcribed, they will be password-protected and stored online behind the MD Anderson firewall.

## Proprietary of MD Anderson Cancer Center

NCT05308407 April 24, 2025

Up to 80 participants will take part in this study. All will take part at MD Anderson.

#### 4. Provide participant with additional Information

You should discuss the risks of the focus groups with the study chair. The known risks are listed in this form, but they will vary from person to person. Some questions may make you feel upset or uncomfortable. You may refuse to answer any question. If you have concerns after taking part in the focus group, you are encouraged to contact the study chair.

We will use a pseudonym (different name) during the focus groups so that your name will be confidential.

Although every effort will be made to keep study data safe, there is a chance that your personal information could be lost or stolen. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

Your participation or non-participation in this study will not affect your medical care in any way.

If you choose to withdraw from this study your medical care will not be affected. If you choose to withdraw from this study, the data collected about you up until withdrawal can be used and included in data analysis. However, no further information about you will be collected.

Your participation in this study will be complete after you complete the focus group.

This is an investigational study. There will be no cost to you for taking part in this study. You will be compensated with a \$15 gift card for taking part in this study. There are no benefits for you in this study. Your participation is completely voluntary and your responses will be kept confidential. You may choose not to take part in this study.

#### **Describe the Use and Sharing of Protected Health Information**

During the course of this study, the research team at The University of Texas MD Anderson Cancer Center will be collecting information about you that they may share with health authorities, study monitors who check the accuracy of the information, and individuals who put all the study information together in report form. By agreeing to take part in this study, you are providing authorization for the research team to use and share your information at any time. If you do not want to authorize the use and disclosure of your information, you may choose not to take part in this study. There is no expiration date for use of this information. You may withdraw your authorization at any time, in writing, for any reason as long as that information can be connected to you. You can learn more about how to withdraw your authorization by calling the Chief Privacy Officer at 713-745-6636 or by contacting the study chair, Keri Schadler at 713-794-1035 with any questions you have about the

#### NCT05308407 April 24, 2025

# Proprietary of MD Anderson Cancer Center

study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB - a committee that reviews research studies) at 713-792-6477.

### 5. Length of the Study

It will take no more than 2 hours to take part in the focus group. Are you interested in taking part in this study?

Participant's answer:

- Yes (Continue with the next section)
- No (Thank them and document the answer)

### 6. Document Participant Consent

Before you can take part in this study, you must agree to the following statements:

 You have been given the description of the study, and you have decided to take part in the research study described to you. (Yes – No)

| Name of the researcher obtaining the verbal consent/Credentials/Signature/Date |
|---|